CLINICAL TRIAL: NCT00482456
Title: Influence of the MTHFR 677C>T Mutation on Homocysteine Levels After Nitrous Oxide Anesthesia.
Brief Title: Homocysteine After Nitrous Oxide Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EK 286/2004
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Last update posted 2007-06-05 (Estimated); Status verified 2007-05

CONDITIONS: Anesthesia, General; Adverse Effects; Nitrous Oxide
Keywords: Nitrous oxide; Homocysteine; folate; vitamin B12
MeSH Terms: interventions — Nitrous Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nitrous oxide

SUMMARY:
Our study looks at the interaction of a common mutation in the MTHFR gene and the risk of developing higher homocysteine levels after nitrous oxide (N2O) anesthesia.

Specifically, we want to test the hypothesis that healthy patients carrying the MTHFR 677C>T haplotype develop abnormal homocysteine levels after nitrous oxide anesthesia.

DETAILED DESCRIPTION:
Nitrous oxide - laughing gas - is a widely used anaesthetic gas with many favourable but also some dangerous properties. Among the latter is the increase in homocysteine levels after nitrous oxide (N2O) exposure by inhibition of enzymes in the vitamin B12 pathway. Elevated homocysteine levels have been found to be an independent risk factor for ischemic events and are associated with an increased risk for perioperative myocardial ischemia. If a patient carries one or more loss-of-function mutations in enzymes of the methionine/homocysteine/folate pathway he is at an increased risk for hyperhomocysteinemia and if exposed to N2O might suffer severe, sometimes disastrous neurological damage. Recently, a case report in the New England Journal of Medicine reported the death of a child with an enzyme defect in the MTHFR gene after anaesthesia with nitrous oxide (NEJM 2003;349:45-50).

Thus, we are convinced that if we can determine the risk of patients who carry mutations in the MTHFR gene and undergo anaesthesia with N2O for developing pathological levels of homocysteine, we can add an important piece of information to the safety profile of N2O.

Our study tests the hypothesis that patients who carry the 677C<T mutation in the MTHFR gene (the most common mutation) have a higher risk of developing hyperhomocysteinemia after N2O anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for general anaesthesia (> 2 hours)
* Age > 18 years
* ASA status I-II

Exclusion Criteria:

* Pregnancy
* Age < 18 years
* contraindication against N2O: pneumothorax, mechanical bowel obstruction, middle ear occlusion, laparoscopic surgery
* recent use of vitamin preps (B12, B6, folate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2005-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Homocysteine levels dependent on MTHFR genotype | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nagele, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Dept of Anesthesiology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Nagele P, Zeugswetter B, Eberle C, Hupfl M, Mittlbock M, Fodinger M. A common gene variant in methionine synthase reductase is not associated with peak homocysteine concentrations after nitrous oxide anesthesia. Pharmacogenet Genomics. 2009 May;19(5):325-9. doi: 10.1097/FPC.0b013e328328d54c. PMID 19339913
- [Derived] Nagele P, Zeugswetter B, Wiener C, Burger H, Hupfl M, Mittlbock M, Fodinger M. Influence of methylenetetrahydrofolate reductase gene polymorphisms on homocysteine concentrations after nitrous oxide anesthesia. Anesthesiology. 2008 Jul;109(1):36-43. doi: 10.1097/ALN.0b013e318178820b. PMID 18580170